CLINICAL TRIAL: NCT05176171
Title: Advanced Surface Ablation With Corneal Cross Linking in Mild Keratoconus
Brief Title: Surface Ablation With Corneal Cross Linking in Mild Keratoconus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University (Other)
Collaborators: Negah Eye Center (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, farinaz doroodgar, Ophthalmologist, Shahid Beheshti University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBMU
Record Dates: First submitted 2020-04-05; First posted 2022-01-04 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-01

CONDITIONS: Keratoconus; Corneal Cross-Linking
MeSH Terms: conditions — Keratoconus | interventions — Photorefractive Keratectomy; Corneal Cross-Linking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photorefractive Keratectomy with Corneal Cross-Linking (Experimental): For correction of refractive error
  Interventions: Procedure: Photorefractive Keratectomy with Corneal Cross-Linking

INTERVENTIONS:
Procedure: Photorefractive Keratectomy with Corneal Cross-Linking — To our knowledge, this study is one of the first to compare the visual results of non-topography-guided and topography-guided photorefractive keratectomy (PRK) applying sequential and simultaneous corneal cross-linking (CXL) treatment for keratoconus. Considering recent advances in cross-linking and imaging in keratoconus, the outcomes of this study can lead us to several non-invasive algorithm management options.

SUMMARY:
Interventional and comparative prospective study: Sixty-nine eyes (38 patients) suffering from keratoconus (stages 1-2 Amsler-Krumeich classification) will be divided into four groups. The four groups underwent topography- and non-topography-guided PRK with sequential and simultaneous CXL. The main outcome measures will be pre-and postoperative uncorrected distance visual acuity (UDVA), best-corrected distance visual acuity (CDVA), manifest refraction, contrast sensitivity, and keratometry

ELIGIBILITY:
Inclusion criteria for the study focused on patients over 34 (range from 34 to 41) with stable corneal topography and refraction for at least six months and an estimated residual bed thickness of >410 µm.

exclusion from the study included the presence of macular or retinal disease, dry eye, history of recurrent corneal erosions, anterior segment abnormalities, unstable refractive error, post-surgically residual stromal bed thickness of under 350 mm, autoimmune disease, collagen vascular disease, immunosuppressive therapy, or current use of systemic corticosteroids, diabetes mellitus, pregnancy, and lactation.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2023-07-05 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 3 year
  Evaluation of the uncorrected visual acuity, best corrected visual acuity, astigmatism, intraocular pressure and endothelial cell loss before and after the last operation.

CONTACTS AND LOCATIONS:
Overall Officials: Azad sanginabadi, PhD, Principal Investigator — Iran University of Medical Sciences
Locations (1):
- Negah Eye Hospital, Tehran, Iran